CLINICAL TRIAL: NCT04542447
Title: An Open Label Proof of Concept Study to Assess Aspects of Safety and Efficacy of Nuvastatic™ (C5OSEW5050ESA) as an Immunomodulator Adjuvant Therapy to the Standard Care of Treatment in Covid 19 Patients.
Brief Title: To Evaluate Safety and Efficacy of Nuvastatic as an Immunomodulator Adjuvant Therapy in COVID-19 Patients.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Natureceuticals Sdn Bhd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIAG-CSP-037
Record Dates: First submitted 2020-09-06; First posted 2020-09-09 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Immunomodulator in COVID 19, Intervention - Sequentially numbered IP kits
Masking Description: An open label proof of concept study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nuvastatic + standard treatment (Active Comparator): 5 patients, dosage: 3000 mg of Nuvastatic™ (C5OSEW5050ESA) each day plus standard of care thrice daily (morning, afternoon and evening (one sachet each) to be taken for 14 days in Covid-19 patients.
  Interventions: Drug: Nuvastatic
- Placebo (Placebo Comparator): 5 patients, dosage: 3000 mg of placebo each day plus standard of care thrice daily (morning, afternoon and evening (one sachet each) to be taken for 14 days in Covid-19 patients.
  Interventions: Drug: Nuvastatic

INTERVENTIONS:
Drug: Nuvastatic — Polymolecular botanical standardized extract Orthosiphon stamineus/Orthosiphon aristatas as an immunomodulator adjuvant therapy
  Other Names: C5OSEW5050ESA

SUMMARY:
A two arm open label multi-centered randomized interventional trial is proposed to assess aspects of safety and efficacy of Nuvastatic™ (Serial No: C5OSEW5050ESA) . Two parallel groups of (1:1) ratio comparing Nuvastatic™ versus standard care will be conducted on patients on oxygen saturation (SaO2) of 94% or less while they are breathing ambient air or a ratio of the partial pressure of oxygen (Pao2) to the fraction of inspired oxygen (Fio2) (PaO2:FiO2) at or below 300 mg Hg.

Primary Outcome Measures: time to clinical improvement, defined as the time from randomization to an improvement of two points (from the status at randomization) on a seven-category ordinal scale or live discharge from the hospital, whichever comes first.

Secondary Outcome Measures: Clinical status as assessed with the seven-category ordinal scale on days 7 and 14, mortality at day 28.

1. The duration of mechanical ventilation.
2. The duration of hospitalization in survivors.
3. The time (in days) from treatment initiation to death.
4. Virologic measures included the proportions with viral RNA detection over time and viral RNA titer area under-curve (auc) measurements.

DETAILED DESCRIPTION:
This study will propose Nuvastiatic™ as a new lead therapeutic agent for SARS-CoV-2, and new insights for currently ongoing clinical trials to treat SARS-CoV-2 infections. Nuvastatic™ could be used as potential anti-coronavirus therapy that acts on the human immune system or human cells as an immune modulator, and the other on coronavirus itself as an antiviral agent. In terms of the human immune system, the innate immune system response plays an important role in controlling the replication and infection of coronavirus, and interferon gamma, interleukins, Th cells, granulocyte macrophage are expected to enhance the immune response.

ELIGIBILITY:
Inclusion Criteria:

1. Male and nonpregnant female patients 18 years of age or older eligible if they had a diagnostic specimen that was positive on RT-PCR. -
2. For Mild - Moderate cases: Subjects who show positive for nasal swab test at screening using RT-PCR protocol for Covid 19.
3. For Severe cases - Has an oxygen saturation (Sao2) of 94% or less while they are breathing ambient air or a ratio of the partial pressure of oxygen (Pao2) to the fraction of inspired oxygen (Fio2) (Pao2:Fio2) at or below 300 mg Hg.
4. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Female subjects who are pregnant or breastfeeding.
2. Patients who are allergic to this medicine
3. Patients allergic to content of study product
4. Patients with diabetes.
5. Patients accompanied by serious physical diseases of heart, lung, brain, etc.
6. Patients have any condition that in the judgement of the Investigators would make the subject inappropriate for entry into this study.
7. Patients who are not able to take drugs orally.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate safety and efficacy Nuvastatic™ (C5OSEW5050ESA) | 14 Days
  Time to clinical improvement, defined as the time from randomization to an improvement of two points (from the status at randomization) on a seven-category ordinal scale or live discharge from the hospital, whichever comes first.
IL-6 reduction | 14 Days
  Improvement of Biomarkers: IL-6 reduction
Serum c-reactive protein (CRP) | 14 Days
  Improvement of Biomarkers:key inflammatory markers Serum c-reactive protein (CRP)
IgG | 14 Days
  Improvement of Biomarkers:key inflammatory markers IgG
Hb | 14 Days
  Improvement of Biomarkers:key inflammatory markers Hb
Total leucocyte count | 14 Days
  Improvement of Biomarkers:key inflammatory markers Total leucocyte count
F2-Isoprostane | 14 Days
  Improvement of Biomarkers:key inflammatory markers urinary F2-Isoprostane.
Improvement in ARDS associated clinical symptoms cause | 14 Days
  Role of VEGF as potential therapeutic target in acute respiratory distress syndrome (ARDS)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Vinaik, Principal Investigator — Navin Hospital
Locations (1):
- Navin Hospital, Ghaziabad, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No
Institutional sharing